CLINICAL TRIAL: NCT07083180
Title: Effectiveness of Medical Hypnosis in Virtual Reality on Preoperative Anxiety in Carpal Tunnel Surgery Interventional Study With Minimal Risks and Constraints, Single-center, Prospective
Brief Title: Effectiveness of Medical Hypnosis in Virtual Reality on Preoperative Anxiety in Carpal Tunnel Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique MEGIVAL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-26-MEG
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Patients are invited to practice a recreational activity to reduce pre-operative anxiety
  Interventions: Other: Recreative activity
- Virtual hypnosis arm (Experimental): patients undergoing medical hypnosis using virtual reality
  Interventions: Other: Medical Hypnosis by virtual reality

INTERVENTIONS:
Other: Recreative activity — Patients practice a leisure activity before surgery (20 minutes)
  Arms: Control arm
Other: Medical Hypnosis by virtual reality — Patients benefit from a medical hypnosis session using virtual reality (20 minutes)
  Arms: Virtual hypnosis arm

SUMMARY:
Anxiety is a predominant factor among patients prior to surgery, particularly in the context of outpatient surgery, where the speed of care and same-day discharge can exacerbate this stress. National patient satisfaction surveys, such as e-SATIS CA, show that many patients report significant anxiety before their surgery, which can affect the outcome of the operation and the recovery process. Medical hypnosis has been shown to be an effective way to reduce anxiety in patients before surgery. Indeed, several studies highlight the psychological and physiological benefits of this method for patients who are anxious before minor or major surgery. Hypnosis allows for deep relaxation, helping to better manage the emotions and fears associated with surgery. New technologies, such as virtual reality, are now being integrated into hypnosis practices to improve their effectiveness. Virtual immersion provides distraction and an environment conducive to hypnosis, facilitating induction and further reducing preoperative anxiety. In this context, we wish to conduct a single-center clinical investigation to determine whether the use of the HypnoVR virtual reality headset can help reduce anxiety in patients undergoing outpatient carpal tunnel surgery.

ELIGIBILITY:
Inclusion Criteria:

* First surgery of carpal tunnel

Exclusion Criteria:

* Patients undergoing treatment for anxiety
* Uncontrolled epilepsy
* Visual (binocular vision) and/or hearing impairments preventing the use of virtual reality
* Pregnancy / breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Anxiety level | 15 minutes before leisure activity or virtual reality session ; 15 minutes after leisure activity or virtual reality session
  Anxiety level will be measured before and after intervention, using STAI-state Anxiety scale (20 questions with 4 points Likert scale from "not at all" to "totally")

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique MEGIVAL, Saint-Aubin-sur-Scie, France

IPD SHARING:
Plan to Share IPD: No